CLINICAL TRIAL: NCT00467857
Title: A Randomized, Controlled, Parallel Group, Multi-center, Open Label Study Comparing Common Surgical Skin Preparation Solutions in Combination With InteguSeal Versus Common Surgical Skin Preparation Solutions to Reduce Skin Flora Contamination.
Brief Title: Study of the Combination of a Cyanoacrylate and Surgical Solutions in Reducing Skin Flora Contamination
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kimberly-Clark Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IS 100-06-0001
Record Dates: First submitted 2007-04-27; First posted 2007-05-01 (Estimated); Results first posted 2011-02-11 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2011-01

CONDITIONS: Skin Flora Contamination
Keywords: cyanoacrylates; microbial sealants; skin flora contamination; surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- InteguSeal* and standard surgical preparation solutions (Active Comparator): InteguSeal* microbial skin sealant was applied to surgical sites prior to incision after standard surgical skin preparation in patients undergoing coronary artery bypass graft (CABG) surgery
  Interventions: Procedure: InteguSeal* skin sealant and standard surgical preparation
- Standard surgical skin preparation alone (Other): Prior to incision, standard surgical skin preparation in patients undergoing coronary artery bypass graft (CABG) surgery
  Interventions: Other: Standard preoperative skin preparation

INTERVENTIONS:
Procedure: InteguSeal* skin sealant and standard surgical preparation — Surgical skin preparation prior to incision using InteguSeal* skin sealant following standard surgical preparation with povidone iodine or 0.7% available iodine in isopropyl alcohol 74% w/w.
  Other Names: Kimberly Clark InteguSeal* Microbial Sealant
  Arms: InteguSeal* and standard surgical preparation solutions
Other: Standard preoperative skin preparation — Surgical skin preparation prior to incision using standard surgical preparation with povidone iodine or 0.7% available iodine in isopropyl alcohol 74% w/w.
  Arms: Standard surgical skin preparation alone

SUMMARY:
The purpose of this study is to determine if there is a qualitative reduction in microbial skin flora post-surgery compared to pre-surgery when a cyanoacrylate based microbial sealant is used in combination with a surgical skin preparation solution.

DETAILED DESCRIPTION:
The CDC states that there are two sources of surgical site infection (SSI) pathogens- endogenous and exogenous. The endogenous flora of the patient's skin, mucous membranes, or hollow viscera are the source of pathogens for most SSIs. In addition to the known sources of SSI pathogen, there are also known risk factors for SSI. The risk factors for SSIs may be patient-related, or related to the preoperative, intra-operative, and post-operative surgical treatment and care of the patient. Many known risk factors that contribute to SSIs include, but are not limited to age, nutritional status, co-morbidities, length of pre-operative stay, duration of operation, preoperative skin prep, and surgical techniques. In addition, there are certain surgical procedures in which the risks for developing SSI are greater than other surgical procedures. While there are various pre-operative and post-operative techniques or approaches to prevent these infections in patients undergoing surgeries, such as pre-operative skin care techniques, appropriate use of antibiotic prophylaxis, and the use of other post-operative anti-microbial methods, by immobilizing the patient's endogenous skin flora, an opportunity exists to reduce the rate of skin flora contamination which leads to wound contamination.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for an elective Coronary Artery Bypass Graft (CABG) surgical procedure with median sternotomy utilizing either the saphenous vein and/or radial artery as one of the graft sites within 28 days of the screening date, as documented by a Cardiothoracic Surgeon who is the Principal Investigator or sub-investigator. This includes subjects who are also receiving internal mammary artery grafts in addition to saphenous vein and/or radial artery grafts.
* The skin near or around the proposed incision sites should be intact.

Exclusion Criteria:

* Known sensitivity or allergy to cyanoacrylate, isopropyl alcohol, iodine or iodine-containing products or tape allergies.
* Female subjects that are nursing or actively lactating.
* Abnormal skin condition adjacent to or at the surgical incision sites.
* Hair removal at the surgical sites prior to entrance to the operating suite.
* Use of antimicrobial impregnated incise drapes (i.e. Ioban®).
* Hospital stay of >14 days immediately prior to scheduled CABG surgery.
* Use of chemotherapy agents, within 30 days prior to Visit 1 screening.
* Scheduled for additional chemotherapy for the duration of the study.
* Known positive Human Immunodeficiency Virus (HIV) with a CD4 count < 350 mm3. If HIV status is not known, the subject is not excluded.
* Currently taking antibiotics for an infection (within 30 days prior to Visit 1).
* Has had therapeutic radiation to the chest within 30 days of visit 1. This does not include subjects who receive chest xrays.
* Pre-operatively scheduled to have concomitant procedures with coronary artery bypass graft procedure.
* Scheduled to receive only one incision (a median sternotomy) without a planned saphenous vein graft and/or a radial artery graft donor site.
* Renal dialysis currently or within 30 days of visit 1.
* Morbid Obesity (Subjects with a Body Mass Index (BMI) > 37).
* Neutropenia (absolute neutrophil count <1000/mm3).
* Pre-operatively on an intra-aortic balloon pump or mechanical assist device.
* Has received an experimental drug or used an experimental medical device within 30 days prior to Visit 1.
* Employees of the investigator or study center with direct involvement in the proposed study or other studies under the direction of that investigator or study center.
* Any condition, which in the opinion of the investigator would exclude the subject from the study.
* Patients on steroid use for more than 1 week within 30 days of visit 1.
* Patients on immunosuppressive therapy within 30 days of visit 1.
* Depilatory creams with containing antibiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2007-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte D Owens, MD, Study Director — Kimberly-Clark Corporation
Locations (5):
- Wellstar Health Systems, Marietta, Georgia, United States
- Heart Institute- Dept of Thoracic Surgery, São Paulo, São Paulo, Brazil
- Hospital Dr. Hernan Henriquez Aravena, Temuco, Chile
- Charité, Humboldt University- Department of Cardiovascular Surgery, Berlin, Germany
- National Heart Centre, Singapore, Singapore

REFERENCES:
- [Background] Dohmen PM. Influence of skin flora and preventive measures on surgical site infection during cardiac surgery. Surg Infect (Larchmt). 2006;7 Suppl 1:S13-7. doi: 10.1089/sur.2006.7.s1-13. PMID 16834542
- [Background] Malangoni MA, Cheadle WG, Dodson TF, Dohmen PM, Jones D, Katariya K, Kolvekar S, Urban JA. New opportunities for reducing risk of surgical site infection. Roundtable discussion. Surg Infect (Larchmt). 2006;7 Suppl 1:S23-39. doi: 10.1089/sur.2006.7.s1-23. No abstract available. PMID 16834544
- [Background] Fernandez-Ayala M, Nan DN, Farinas-Alvarez C, Revuelta JM, Gonzalez-Macias J, Farinas MC. Surgical site infection during hospitalization and after discharge in patients who have undergone cardiac surgery. Infect Control Hosp Epidemiol. 2006 Jan;27(1):85-8. doi: 10.1086/500334. Epub 2006 Jan 6. PMID 16418996
- [Background] Mangram AJ, Horan TC, Pearson ML, Silver LC, Jarvis WR. Guideline for Prevention of Surgical Site Infection, 1999. Centers for Disease Control and Prevention (CDC) Hospital Infection Control Practices Advisory Committee. Am J Infect Control. 1999 Apr;27(2):97-132; quiz 133-4; discussion 96. PMID 10196487
- [Background] Mertz PM, Davis SC, Cazzaniga AL, Drosou A, Eaglstein WH. Barrier and antibacterial properties of 2-octyl cyanoacrylate-derived wound treatment films. J Cutan Med Surg. 2003 Jan-Feb;7(1):1-6. doi: 10.1007/s10227-002-1154-6. Epub 2002 Oct 9. PMID 12362261
- [Derived] von Eckardstein AS, Lim CH, Dohmen PM, Pego-Fernandes PM, Cooper WA, Oslund SG, Kelley EL. A randomized trial of a skin sealant to reduce the risk of incision contamination in cardiac surgery. Ann Thorac Surg. 2011 Aug;92(2):632-7. doi: 10.1016/j.athoracsur.2011.03.132. Epub 2011 Jun 24. PMID 21704290

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between April 2006 and February 2009 at 5 centers in the United States, Europe, Asia, and Latin America.
Pre-assignment Details: Of 300 patients assessed for eligibility, 7 were not allocated to treatment due to inclusion or exclusion criteria.
Groups:
- InteguSeal* and Standard Surgical Preparation Solutions: Prior to incision, surgical sites were prepared using InteguSeal* following standard surgical preparation with povidone iodine or 0.7% available iodine in isopropyl alcohol 74% w/w. InteguSeal* is a film-forming cyanoacrylate-based microbial skin sealant developed to decrease wound contamination by endogenous skin flora.
- Standard Surgical Preparation Solutions: Prior to incision, standard surgical preparation with povidone iodine or 0.7% available iodine in isopropyl alcohol 74% w/w.
Period: Overall Study
Arm/Group | InteguSeal* and Standard Surgical Preparation Solutions | Standard Surgical Preparation Solutions
Started | 146 | 147
Completed | 143 | 139
Not Completed | 3 | 8
Not completed — Adverse Event | 1 | 0
Not completed — Withdrew consent | 2 | 0
Not completed — Death | 0 | 1
Not completed — Discharged from court service | 0 | 1
Not completed — Emergency care required | 0 | 1
Not completed — Did not meet inclusion/exclusion criteri | 0 | 2
Not completed — Discontinuation reason missing | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | InteguSeal* and Standard Surgical Preparation Solutions | Standard Surgical Preparation Solutions | Total
Number analyzed (Participants) | 146 | 147 | 293
Age Continuous [Mean (Standard Deviation); unit: years] | 63.18 (8.53) | 62.94 (9.97) | 63.06 (9.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 18 | 44
  Male | 120 | 129 | 249
Height [Mean (Standard Deviation); unit: meters] — Data for n=145 microbial skin sealant, n=147 control
  meters | 1.67 (0.10) | 1.66 (0.09) | 1.67 (0.10)
Weight [Mean (Standard Deviation); unit: kilograms] | 76.2 (14.4) | 73.8 (12.0) | 75.0 (13.3)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Results for n=145 microbial skin sealant, n=147 control.
  kg/m^2 | 27.3 (4.0) | 26.6 (3.4) | 26.9 (3.71)
Obesity [Number; unit: participants]
  Obese (BMI>30.0 kg/m^2) | 40 | 20 | 60
  Not obese | 106 | 127 | 233
Diabetes mellitus, type 1 or 2 [Number; unit: participants]
  present | 49 | 49 | 98
  absent | 97 | 98 | 195
Tobacco Use [Number; unit: participants]
  yes | 84 | 91 | 175
  no | 62 | 56 | 118
Alcohol Use [Number; unit: participants]
  Yes | 42 | 52 | 94
  No | 104 | 95 | 199
New York Heart Association (NYHA) Functional Classification [Number; unit: participants] — The NYHA Functional Classification provides a simple way of classifying the extent of heart failure. It places patients in one of four categories based on how much they are limited during physical activity:
  Class I: No symptoms and no limitation in ordinary physical activity.
  Class II: Mild symptoms and slight limitation during ordinary activity. Comfortable at rest.
  Class III: Marked limitation in activity due to symptoms, even during less-than-ordinary activity. Comfortable only at rest.
  Class IV: Severe limitations. Experiences symptoms even while at rest.
  participants
    Class I | 29 | 38 | 67
    Class II | 73 | 61 | 134
    Class III | 39 | 43 | 82
    Class IV | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Unique Bacterial Isolates From Pre-skin Preparation to Post-CABG - Sternal Site
Description: Number of unique bacterial colony types isolated from samples of skin flora taken from the sternal incision site after surgery minus before surgery (prior to skin prep). Unique colonies were determined based on Gram stain, colony morphology, catalase, coagulase, or staphylococci latex agglutination and oxidase tests.
Time Frame: Before surgery (prior to skin preparation) and after surgery (after closing fascia)
Population: Per protocol
Measure: Mean (Standard Deviation); unit: isolates
Arm/Group | InteguSeal* and Standard Surgical Preparation Solutions | Standard Surgical Preparation Solutions
Number analyzed (Participants) | 116 | 127
isolates | -1.34 (1.0) | -1.31 (1.0)
Statistical Analysis 1: Comparison: InteguSeal* and Standard Surgical Preparation Solutions vs Standard Surgical Preparation Solutions; The sample size determination was selected to achieve 80% power to detect an absolute 10% difference between the two treatment groups in proportion of qualitative reduction in representative skin flora, at a significance level (alpha) of 0.05 using a two-sided z-test with continuity correction; Test type: Superiority or Other; p = 0.655, Wilcoxon-Rank Sum Test

2. Secondary Outcome: Change in Bacterial Count From Pre-skin Preparation to Post-CABG - Sternal Site
Description: Total bacterial counts from samples of skin flora from the sternal incision site after surgery minus before surgery (prior to skin prep).
Time Frame: Before surgery (prior to skin preparation) and after surgery (after closing fascia)
Population: Per protocol
Measure: Mean (Standard Deviation); unit: log CFU/mL
Arm/Group | InteguSeal* and Standard Surgical Preparation Solutions | Standard Surgical Preparation Solutions
Number analyzed (Participants) | 120 | 131
log CFU/mL | -2.14 (1.4) | -1.99 (1.3)
Statistical Analysis 1: Comparison: InteguSeal* and Standard Surgical Preparation Solutions vs Standard Surgical Preparation Solutions; Test type: Superiority or Other; p = 0.276, Wilcoxon-Rank Sum Test

3. Secondary Outcome: Change in Bacterial Count From Pre-skin Preparation to Post-CABG - Graft Site
Description: Total bacterial counts from samples of skin flora from the graft incision site after surgery minus before surgery (prior to skin prep).
Time Frame: Before surgery (prior to skin preparation) and after surgery (after closing fascia)
Population: Per protocol
Measure: Mean (Standard Deviation); unit: log CFU/mL
Arm/Group | InteguSeal* and Standard Surgical Preparation Solutions | Standard Surgical Preparation Solutions
Number analyzed (Participants) | 119 | 126
log CFU/mL | -2.42 (1.3) | -2.31 (1.2)
Statistical Analysis 1: Comparison: InteguSeal* and Standard Surgical Preparation Solutions vs Standard Surgical Preparation Solutions; Test type: Superiority or Other; p = 0.375, Wilcoxon-Rank Sum Test

4. Secondary Outcome: Post-CABG Procedure Bacterial Count - Sternal Site
Description: Total bacterial counts from samples of skin flora of the sternal incision site taken immediately following the CABG procedure.
Time Frame: Post-surgery
Population: Per protocol
Measure: Mean (Standard Deviation); unit: log CFU/mL
Arm/Group | InteguSeal* and Standard Surgical Preparation Solutions | Standard Surgical Preparation Solutions
Number analyzed (Participants) | 120 | 132
log CFU/mL | 0.58 (1.0) | 0.83 (1.1)
Statistical Analysis 1: Comparison: InteguSeal* and Standard Surgical Preparation Solutions vs Standard Surgical Preparation Solutions; Test type: Superiority or Other; p = 0.039, Wilcoxon-Rank Sum Test

5. Secondary Outcome: Post-CABG Procedure Bacterial Count - Graft Site
Description: Total bacterial counts from samples of skin flora of the graft incision site taken immediately following the CABG procedure.
Time Frame: Post-surgery
Population: Per protocol
Measure: Mean (Standard Deviation); unit: log CFU/mL
Arm/Group | InteguSeal* and Standard Surgical Preparation Solutions | Standard Surgical Preparation Solutions
Number analyzed (Participants) | 119 | 127
log CFU/mL | 0.19 (0.5) | 0.34 (0.7)
Statistical Analysis 1: Comparison: InteguSeal* and Standard Surgical Preparation Solutions vs Standard Surgical Preparation Solutions; Test type: Superiority or Other; p = 0.057, Wilcoxon-Rank Sum Test

6. Secondary Outcome: Change in the Number of Unique Bacterial Isolates From Pre-skin Preparation to Post-incision - Sternal Site
Description: Number of unique bacterial colony types isolated from samples of skin flora from the sternal incision site immediately after the incision minus before surgery (prior to surgical skin prep). Unique colonies were determined based on Gram stain, colony morphology, catalase, coagulase, or staphylococci latex agglutination and oxidase tests.
Time Frame: Before surgery (prior to skin preparation) and immediately after incision
Population: Per protocol
Measure: Mean (Standard Deviation); unit: isolates
Arm/Group | InteguSeal* and Standard Surgical Preparation Solutions | Standard Surgical Preparation Solutions
Number analyzed (Participants) | 116 | 127
isolates | -1.53 (0.9) | -1.59 (1.0)
Statistical Analysis 1: Comparison: InteguSeal* and Standard Surgical Preparation Solutions vs Standard Surgical Preparation Solutions; Test type: Superiority or Other; p = 0.646, Wilcoxon-Rank Sum Test

7. Secondary Outcome: Change in the Number of Unique Bacterial Isolates From Pre-skin Preparation to Post-incision - Graft Site
Description: Number of unique bacterial colony types isolated from samples of skin flora from the graft incision site immediately after the incision minus before surgery (prior to surgical skin prep). Unique colonies were determined based on Gram stain, colony morphology, catalase, coagulase, or staphylococci latex agglutination and oxidase tests.
Time Frame: Before surgery (prior to skin preparation) and immediately after incision
Population: Per protocol
Measure: Mean (Standard Deviation); unit: isolates
Arm/Group | InteguSeal* and Standard Surgical Preparation Solutions | Standard Surgical Preparation Solutions
Number analyzed (Participants) | 118 | 126
isolates | -1.95 (1.1) | -1.98 (1.0)
Statistical Analysis 1: Comparison: InteguSeal* and Standard Surgical Preparation Solutions vs Standard Surgical Preparation Solutions; Test type: Superiority or Other; p = 0.788, Wilcoxon-Rank Sum Test

8. Secondary Outcome: Change in Bacterial Count From Pre-skin Preparation to Post-incision - Sternal Site
Description: Total bacterial counts from samples of skin flora from the sternal incision site immediately after incision minus before surgery (prior to skin prep)
Time Frame: Before surgery (prior to skin preparation) and immediately after incision
Population: Per protocol
Measure: Mean (Standard Deviation); unit: log CFU/mL
Arm/Group | InteguSeal* and Standard Surgical Preparation Solutions | Standard Surgical Preparation Solutions
Number analyzed (Participants) | 120 | 131
log CFU/mL | -2.51 (1.3) | -2.54 (1.2)
Statistical Analysis 1: Comparison: InteguSeal* and Standard Surgical Preparation Solutions vs Standard Surgical Preparation Solutions; Test type: Superiority or Other; p = 0.960, Wilcoxon-Rank Sum Test

9. Primary Outcome: Change in Number of Unique Bacterial Isolates From Pre-skin Preparation to Post-CABG - Graft Site
Description: Number of unique bacterial colony types isolated from samples of skin flora taken from the graft incision site after surgery minus before surgery (prior to skin prep). Unique colonies were determined based on Gram stain, colony morphology, catalase, coagulase, or staphylococci latex agglutination and oxidase tests.
Time Frame: Before surgery (prior to skin preparation) and after surgery (after closing fascia)
Population: Per protocol
Measure: Mean (Standard Deviation); unit: isolates
Arm/Group | InteguSeal* and Standard Surgical Preparation Solutions | Standard Surgical Preparation Solutions
Number analyzed (Participants) | 118 | 126
isolates | -1.88 (1.1) | -1.75 (1.0)
Statistical Analysis 1: Comparison: InteguSeal* and Standard Surgical Preparation Solutions vs Standard Surgical Preparation Solutions; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.359, Wilcoxon-Rank Sum Test

10. Secondary Outcome: Change in Bacterial Count From Pre-skin Preparation to Post-incision - Graft Site
Description: Total bacterial counts from samples of skin flora from the graft incision site immediately after incision minus before surgery (prior to skin prep)
Time Frame: Before surgery (prior to skin preparation) and immediately after incision
Population: Per protocol
Measure: Mean (Standard Deviation); unit: log CFU/mL
Arm/Group | InteguSeal* and Standard Surgical Preparation Solutions | Standard Surgical Preparation Solutions
Number analyzed (Participants) | 119 | 126
log CFU/mL | -2.51 (1.3) | -2.58 (1.2)
Statistical Analysis 1: Comparison: InteguSeal* and Standard Surgical Preparation Solutions vs Standard Surgical Preparation Solutions; Test type: Superiority or Other; p = 0.730, Wilcoxon-Rank Sum Test

11. Secondary Outcome: Post-incision Bacterial Count - Sternal Site
Description: Total bacterial counts from samples of skin flora of the sternal incision site taken immediately following the surgical incision
Time Frame: Immediately after surgical incision
Population: Per protocol
Measure: Mean (Standard Deviation); unit: log CFU/mL
Arm/Group | InteguSeal* and Standard Surgical Preparation Solutions | Standard Surgical Preparation Solutions
Number analyzed (Participants) | 120 | 132
log CFU/mL | 0.21 (0.7) | 0.26 (0.7)
Statistical Analysis 1: Comparison: InteguSeal* and Standard Surgical Preparation Solutions vs Standard Surgical Preparation Solutions; Test type: Superiority or Other; p = 0.348, Wilcoxon-Rank Sum Test

12. Secondary Outcome: Post-incision Bacterial Count - Graft Site
Description: Total bacterial counts from samples of skin flora of the graft incision site taken immediately following the surgical incision
Time Frame: Immediately after surgical incision
Population: Per protocol
Measure: Mean (Standard Deviation); unit: log CFU/mL
Arm/Group | InteguSeal* and Standard Surgical Preparation Solutions | Standard Surgical Preparation Solutions
Number analyzed (Participants) | 119 | 127
log CFU/mL | 0.10 (0.4) | 0.08 (0.4)
Statistical Analysis 1: Comparison: InteguSeal* and Standard Surgical Preparation Solutions vs Standard Surgical Preparation Solutions; Test type: Superiority or Other; p = 0.512, Wilcoxon-Rank Sum Test

13. Secondary Outcome: Number of Patients With SSI at the Sternal Site and/or Graft Site
Description: Number of patients who develop at least one surgical site infection at the sternal or graft site during the 30 day post-op follow-up period
Time Frame: 30 days
Population: Intention to treat
Measure: Number; unit: Participants
Arm/Group | InteguSeal* and Standard Surgical Preparation Solutions | Standard Surgical Preparation Solutions
Number analyzed (Participants) | 146 | 147
Participants | 9 | 14
Statistical Analysis 1: Comparison: InteguSeal* and Standard Surgical Preparation Solutions vs Standard Surgical Preparation Solutions; Test type: Superiority or Other; p = 0.285, Chi-squared

14. Secondary Outcome: Number of Patients With Alcohol Use, Tobacco Use, or Obesity With Surgical Site Infection (SSI)
Description: Number of patients with risk factors of alcohol use, tobacco use, or obesity who developed an SSI at the sternal and/or graft site
Time Frame: 30 days
Population: Subset of Intention to treat participants with alcohol use, tobacco use, or obesity
Measure: Number; unit: Participants
Arm/Group | InteguSeal* and Standard Surgical Preparation Solutions | Standard Surgical Preparation Solutions
Number analyzed (Participants) | 108 | 112
Participants | 5 | 11
Statistical Analysis 1: Comparison: InteguSeal* and Standard Surgical Preparation Solutions vs Standard Surgical Preparation Solutions; Test type: Superiority or Other; p = 0.024, Fisher Exact

ADVERSE EVENTS:
Time Frame: 30 days
Description: Investigators assessed patients for the occurrence of adverse events at each study visit and recorded in case report form. Device-related adverse events, surgical site infections, and death were the only types of adverse events collected.
Arm/Group | InteguSeal* and Standard Surgical Preparation Solutions | Standard Surgical Preparation Solutions
Serious Adverse Events (participants affected / at risk) | 6/146 | 8/147
Other Adverse Events (participants affected / at risk) | 6/146 | 10/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | InteguSeal* and Standard Surgical Preparation Solutions (N=146) | Standard Surgical Preparation Solutions (N=147)
Death (General disorders) | 0 | 3
Sudden death (General disorders) | 1 | 0
Incision site infection (Infections and infestations) | 3 | 2
Mediastinitis (Infections and infestations) | 2 | 2
Osteomyelitis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Hospitalisation (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | InteguSeal* and Standard Surgical Preparation Solutions (N=146) | Standard Surgical Preparation Solutions (N=147)
Arteriovenous graft site infection (Infections and infestations) | 1 | 0
Incision site infection (Infections and infestations) | 3 | 8
Mediastinitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1
Skin graft infection (Infections and infestations) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All publications and presentations resulting from this multi-center trial sponsored by Kimberly-Clark must be approved by all investigators and the sponsor.